CLINICAL TRIAL: NCT07216313
Title: A Phase 1, Open-Label Study to Evaluate the Mutual Drug-Drug Interaction Potential Between Denifanstat and Resmetirom in Healthy Adult Participants
Brief Title: A Drug-Drug Interaction Study of Denifanstat and Resmetirom in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sagimet Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SB2640-CLIN-013
Record Dates: First submitted 2025-10-08; First posted 2025-10-14 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — resmetirom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Effect of resmetirom on pharmacokinetics of denifanstat
  Interventions: Drug: Denifanstat; Drug: Resmetirom
- Cohort 2 (Experimental): Effect of denifanstat on pharmacokinetics of resmetirom
  Interventions: Drug: Denifanstat; Drug: Resmetirom

INTERVENTIONS:
Drug: Denifanstat — Once daily
Drug: Resmetirom — Once daily

SUMMARY:
This is an open-label, 2-cohort study to evaluate the mutual DDI potential between denifanstat and resmetirom in healthy adult participants.

ELIGIBILITY:
Additional inclusion and exclusion criteria may apply.

Inclusion Criteria:

* Seated blood pressure is ≥ 90/40 mmHg and ≤ 140/90 mmHg at the screening visit.
* Seated pulse rate is ≥ 40 bpm and ≤ 99 bpm at the screening visit.
* QTcF interval is ≤ 460 msec (males) and ≤ 470 msec (females) and has ECG findings considered normal or not clinically significant by the PI or designee at the screening visit.
* Liver function test including ALT, AST, ALP and total bilirubin ≤ upper limit of normal at the screening visit.
* Estimated CrCL ≥ 80 mL/min at the screening visit.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (cholecystectomy will not be allowed; uncomplicated appendectomy and hernia repair will be allowed).
* Presence of any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines.
* History or presence of hepatobiliary or thyroid-related disease.
* Significant change (approximately 10% increase or decrease) in weight within 3 months prior to first dosing in the opinion of the PI or designee.
* History of alcoholism or drug/chemical abuse within 2 years prior to check-in.
* Positive results for HIV, HBsAg, or HCV at the screening visit.
* Poor peripheral venous access.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-09-30 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2025-10-20 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve during a dosing interval (tau) at steady state (AUC0-tau) | 7 days
Maximum observed concentration at steady-state (Cmax,ss) | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No